CLINICAL TRIAL: NCT03793478
Title: A Phase 1/2, Multicenter, Dose-Escalating Study To Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy Of Quizartinib Administered in Combination With Re-Induction Chemotherapy, and as a Single-Agent Continuation Therapy, in Pediatric Relapsed/Refractory AML Subjects Aged 1 Month to <18 Years (and Young Adults Aged up to 21 Years) With FLT3-ITD Mutations
Brief Title: Safety and Efficacy of Quizartinib in Children and Young Adults With Acute Myeloid Leukemia (AML), a Cancer of the Blood
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Innovative Therapies For Children with Cancer Consortium (Other); Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AC220-A-U202; 2016-002919-18 (EudraCT Number)
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia recurrent; Relapsed or refractory; FMS-like tyrosine kinase 3 positive; Cancer of the blood; AML; FLT3-ITD mutation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — quizartinib; fludarabine; Cytarabine; Etoposide

STUDY DESIGN:
Intervention Model Description: A single group will progress through a multiple phase study design as described in the detailed description.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): All participants will receive re-induction therapy that includes fludarabine and cytarabine in combination with experimental drug quizartinib. For prophylaxis, IT chemotherapy with cytarabine, methotrexate and prednisolone/hydrocortisone will be given prior to or between re-induction cycles. After completing re-induction therapy, eligible participants may also receive optional consolidation chemotherapy which includes cytarabine, etoposide and quizartinib, if HSCT is not available immediately. After completing re-induction or HSCT successfully, eligible participants can go on to receive continuation therapy with quizartinib.
  Interventions: Drug: Quizartinib; Drug: Fludarabine; Drug: Cytarabine; Drug: Intrathecal (IT) triple chemotherapy prophylaxis; Drug: Etoposide

INTERVENTIONS:
Drug: Quizartinib — Administered orally once daily starting on Day 6 and continuing through Day 28;
  Optional low intensity consolidation with chemotherapy:
  Administered orally once daily starting on Day 1 and continuing through Day 28
  Other Names: Quizartinib dihydrochloride; Vanflyta
Drug: Fludarabine — 30 mg/m^2/day IV infusion given over 30 minutes on Days 1 through 5 (administered based on body weight)
Drug: Cytarabine — 2000 mg/m^2/day IV infusion given over 3 hours on Days 1 through 5 (begin 4 hours after the start of fludarabine) (administered in accordance with standard of care);
  Optional high intensity consolidation with chemotherapy and quizartinib:
  500 mg/m^2/day as a continuous 96-hour IV infusion on Days 1 through 4;
  Optional low intensity consolidation with chemotherapy:
  75 mg/m^2/day as once daily subcutaneous or IV on Days 1 through 4 and Days 15 through 18
Drug: Intrathecal (IT) triple chemotherapy prophylaxis — IT cytarabine, methotrexate, and either prednisolone or hydrocortisone; doses are based on the participant's age and standard practice at each site
Drug: Etoposide — Optional high intensity consolidation with chemotherapy and quizartinib:
  100 mg/m^2/dose once daily as an IV infusion over 3 hours on Days 1 through 5

SUMMARY:
Quizartinib is an experimental drug. It is not approved for regular use. It can only be used in medical research.

Children or young adults with a certain kind of blood cancer (FLT3-ITD AML) might be able to join this study if it has come back after remission or is not responding to treatment.

DETAILED DESCRIPTION:
The medical condition being investigated is relapsed or refractory AML in participants aged ≥1 month to ≤21 years with Feline McDonough Sarcoma (FMS)-like tyrosine kinase 3 (FLT3)-internal tandem duplication (ITD) mutations (FLT3-ITD AML), following failure of front-line intensive chemotherapy.

The trial will be conducted in multiple phases. An independent data monitoring committee (DMC) will protect the rights, safety, and well-being of participants by monitoring the progress and results. The DMC will comprise qualified physicians and scientists who are not Investigators in the study and not otherwise directly associated with the Sponsor and will be convened at the end of Phase 1.

A. Dose Escalation/De-escalation Phase:

Number of participants is determined by age group. Participants will be enrolled by dose-level to determine the recommended Phase 2 dose (RP2D) of quizartinib for pediatric participants that provides similar exposure to adult patients treated at the target adult dose of 60 mg orally once daily.

B. Dose-Expansion Phase:

Participants will receive the RP2D of quizartinib for their respective age group.

During both dose escalation and dose expansion phases, participants will receive:

Re-Induction Therapy

* Intrathecal (IT) triple chemotherapy prophylaxis prior to and between cycles
* In re-induction Cycles 1 and 2, fludarabine/cytarabine (FLA) followed by quizartinib as a single agent

Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) Period:

After re-induction therapy, participants will be evaluated for eligibility to undergo allogeneic hematopoietic stem cell transplant (HSCT). Eligible participants may receive a single 28-day cycle of consolidation therapy (standard of care chemotherapy with or without quizartinib) if an allogeneic HSCT is not available immediately. The options for consolidation therapy are as follows:

* High intensity chemotherapy with quizartinib, or
* Low intensity chemotherapy alone, or
* Low intensity therapy with quizartinib as a single agent

Continuation Therapy:

Participants in remission after HSCT, or who are not eligible for HSCT but achieve at least a partial remission (PR) after re-induction, will receive up to 12 continuous 28-day cycles of quizartinib continuation therapy at the same dose received during re-induction in the dose expansion phase.

Long-term Follow-up:

The long-term follow-up phase begins upon completion of 12 cycles of quizartinib Continuation Therapy or permanent discontinuation of quizartinib at any time. After completion of the 30-day safety follow-up visit, subsequent visits will occur at the following frequencies to assess survival and anti-leukemic treatments:

* every 3 months for the first 2 years, and then
* once a year thereafter until the last participant enrolled has been followed for three years from the date of enrollment

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for enrollment into the study:

* Has diagnosis of AML according to the World Health Organization (WHO) 2008 classification with ≥5% blasts in bone marrow, with or without extramedullary disease
* In first relapse or refractory to first-line high-dose chemotherapy with no more than 1 attempt (1 to 2 cycles of induction chemotherapy) at remission induction - prior HSCT is permitted
* Has presence of the FLT3-ITD activating mutation in bone marrow or peripheral blood as defined in the protocol
* Is between 1 month and 21 years of age at the time the Informed Consent/Assent form is signed
* Has protocol-defined adequate performance status score
* Has fully recovered from the acute clinically significant toxicity effects of all prior chemotherapy, immunotherapy, or radiotherapy, per protocol guidelines
* Has protocol-defined adequate renal, hepatic and cardiac functions
* If of reproductive potential, is permanently sterile or agrees to use highly effective birth control upon enrollment, during the period of therapy, and for 6 months following the last dose of quizartinib, etoposide, fludarabine, methotrexate, or cytarabine, whichever is later
* If female of child-bearing potential, tests negative for pregnancy and agrees not to breast feed
* Male participants must be surgically sterile or willing to use highly effective birth control during the treatment period, and for 6 months following the last dose of quizartinib, etoposide, fludarabine, methotrexate, or cytarabine, whichever is later.
* Participant/legal representative is capable of understanding the investigational nature of the study, potential risks, and benefits, and the patient (and/or legal representative) signs a written assent/informed consent

Exclusion Criteria:

Participants who meet any of the following criteria will be disqualified from entering the study:

* Has been diagnosed with isolated central nervous system relapse, acute promyelocytic leukemia (APL), juvenile myelomonocytic leukemia, French-American-British classification M3 or WHO classification of APL with translocation, or with myeloid proliferations related to Down syndrome
* Has uncontrolled or pre-defined significant cardiovascular disease as detailed in the protocol
* Has systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment. The patient must be off vasopressors and have negative blood cultures for at least 48 hours prior to the start of systematic protocol therapy.
* Has known active clinically relevant liver disease (e.g., active hepatitis B or active hepatitis C)
* Has known history of human immunodeficiency virus (HIV)
* Has history of hypersensitivity to any of the study medications or their excipients
* Is receiving or is anticipated to receive concomitant chemotherapy, radiation, or immunotherapy other than as specified in the protocol
* Has any significant concurrent disease, illness, psychiatric disorder or social issue that would compromise subject safety or compliance, interfere with consent/assent, study participation, follow up, or interpretation of study results
* Is currently participating in another investigative interventional procedure (observational or long-term interventional follow-up is allowed)
* Is otherwise considered inappropriate for the study by the Investigator

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of dose-limiting toxicities (Phase 1) | Re-induction Cycle 1 Day 1 up to Day 28 (each cycle is 28 days)
Composite complete remission (CRc) rate among participants with acute myeloid leukemia (AML) (Phase 1 and 2) | within 8 years, 8 months
  CRc rate is defined as percentage of participants with best response of complete remission (CR) or CR with incomplete hematological recovery (CRi) after completion of up to 2 re-induction cycles
Pharmacokinetic parameter area under the concentration curve for quizartinib and AC886 (Phase 1 and 2) | Re-induction Phase 1 and 2,Cycle 1: Days 6, 20:Predose, 1 hour (Phase 1 only), 2, 4, and 6 hours; Days 7 and 21:24 hours; Phase 1 and 2 Cycle 2: Days 6 and 20:predose, 3 hours; Continuation Cycle 1 Days 1 and 15:predose, 2-4 hours (each cycle, 28 days)
Pharmacokinetic parameter apparent clearance (CL/F) for quizartinib and AC886 (Phase 1 and 2) | Re-induction Phase 1 and 2,Cycle 1: Days 6, 20:Predose, 1 hour (Phase 1 only), 2, 4, and 6 hours; Days 7 and 21:24 hours; Phase 1 and 2 Cycle 2: Days 6 and 20:predose, 3 hours; Continuation Cycle 1 Days 1 and 15:predose, 2-4 hours (each cycle, 28 days)
Pharmacokinetic parameter apparent volume of distribution (Vz/F) for quizartinib and AC886 (Phase 1 and 2) | Re-induction Phase 1 and 2,Cycle 1: Days 6, 20:Predose, 1 hour (Phase 1 only), 2, 4, and 6 hours; Days 7 and 21:24 hours; Phase 1 and 2 Cycle 2: Days 6 and 20:predose, 3 hours; Continuation Cycle 1 Days 1 and 15:predose, 2-4 hours (each cycle, 28 days)

SECONDARY OUTCOMES:
Complete remission (CR) rate among participants with AML (Phase 1 and 2) | on Day 56 (± 3 Days) for the last subject, within 4 years
  CR rate is defined as the percentage of participants achieving CR after completion of up to 2 re-induction cycles
Complete remission with incomplete recovery (CRi) rate among participants with AML (Phase 1 and 2) | on Day 56 (± 3 Days) for the last subject, within 4 years
  CRi rate is defined as the percentage of participants achieving CRi after completion of up to 2 re-induction cycles
Duration of CR among participants with AML (Phase 1 and 2) | within 8 years, 8 months
  Duration of CR is defined as the time from the first documented CR until documented relapse
Duration of CRi among participants with AML (Phase 1 and 2) | within 8 years, 8 months
  Duration of CRi is defined as the time from the first documented CRi until documented relapse
Duration of composite complete remission (CRc) among participants with AML (Phase 1 and 2) | within 8 years, 8 months
  Duration of CRc is defined as the time from the first documented CR or CRi until documented relapse
Complete remission (CR) rate after completion of re-induction Cycle 1 among participants with AML (Phase 1 and 2) | on Day 56 (± 3 Days) for the last subject, within 4 years
  CR rate after completion of re-induction Cycle 1 is defined as the percentage of participants achieving a CR after completion of re-induction Cycle 1
Complete remission with incomplete recovery (CRi) rate after completion of re-induction Cycle 1 among participants with AML (Phase 1 and 2) | on Day 56 (± 3 Days) for the last subject, within 4 years
  CRi rate after completion of re-induction Cycle 1 is defined as the percentage of participants achieving a CRi after completion of re-induction Cycle 1
Composite complete remission (CRc) rate after completion of re-induction Cycle 1 among participants with AML (Phase 1 and 2) | on Day 56 (± 3 Days) for the last subject, within 4 years
  CRc rate after completion of re-induction Cycle 1 is defined as the percentage of participants achieving CRc after completion of re-induction Cycle 1
Time to relapse among participants with AML (Phase 1 and 2) | within 8 years, 8 months
  Time to relapse is defined as the time from the first documented response (CR, CRi) until documented relapse
Rate of relapse among participants with AML after 1, 2 and 3 years (Phase 1 and 2) | within 8 years, 8 months
  Rate of relapse is defined as the percentage of participants who achieved CRc at the end of re-induction and had relapsed at 3 categorical time points Categories: 1 year, 2 years, 3 years
Cumulative incidence of relapse among participants with AML at the end of study (Phase 1 and 2) | within 8 years, 8 months
  Cumulative incidence of relapse at the end of the study is defined as the percentage of participants who achieved CRc at the end of re-induction and relapsed by the end of the study
Overall survival among participants with AML at 1, 2, and 3 years (Phase 1 and 2) | within 8 years, 8 months
  Overall survival is defined as the time from the start of re-induction therapy until death from any cause
Event-free survival among participants with AML at 1, 2, and 3 years (Phase 1 and 2) | within 8 years, 8 months
  Event-free survival is defined as the time from the start of re-induction therapy until the earliest date of the following:
  * Refractory disease at the end of re-induction
  * Relapse after CR or CRi
  * Death from any cause at any time during the study
Number of participants proceeding to high-dose conditioning therapy/allogeneic hematopoietic stem cell transplantation (HSCT) (including transplant-related mortality) among participants with AML (Phase 1 and 2) | within 8 years, 8 months
Rate of CRc (CR or CRi) without minimal residual disease (MRD) using next generation sequencing among participants with AML (Phase 1 and 2) | within 8 years, 8 months
  MRD is defined as the presence of leukemic cells in the bone marrow detected above a predefined cut-off level by a validated assay in participants who achieved a CR or CRi
  Categories: at screening, at re-induction cycle 1, at re-induction cycle 2, at time of relapse
Acceptability of including the palatability of quizartinib formulations among participants with AML (Phase 1 and 2) | within 8 years, 8 months
  Acceptability is assessed by palatability using a 5-point hedonic scale (from "Super bad" to "Super good") for participants who are developmentally able to answer. If unable, the caregiver provides information in a free text field stating whether the participant spit it out, may not have liked the flavor, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (27):
- United States (11):
  - Loma Linda University Cancer Center, Loma Linda, California
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - A.I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - The University of Texas Southwestern Medical Center Children's Health, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - British Columbia Children's Hospital, Vancouver
- Rigshospitalet, Copenhagen, Denmark
- France (3):
  - Centre Léon Bérard, Lyon
  - Hôpital Armand-Trousseau, Paris
  - Hôpital des Enfants, Toulouse
- Israel (2):
  - Rambam Medical Center, Haifa
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (3):
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - IRCCS Ospedale Pediatrico Bambino Gesù, Rome
  - Ospedale Infantile Regina Margherita, Torino
- Prinses Maxima Centrum voor Kinderoncologie, Utrecht, Netherlands
- Spain (2):
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario La Paz, Madrid
- Sahlgrenska Universitetssjukhuset - Drottning Silvias Barn- och Ungdomssjukhus, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/